CLINICAL TRIAL: NCT03115060
Title: Comparison of Plasmalyte A, Normal Saline and Ringer Lactate as Intraoperative Fluids in Patients Undergoing Renal Transplantation.
Brief Title: Comparison of Plasmalyte A, Normal Saline and Ringer Lactate as Intraoperative Fluid During Renal Transplantation
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Post Graduate Institute of Medical Education and Research, Chandigarh (Other)
Responsible Party: Principal Investigator, Dr Vikas Saini, Associate Professor, Post Graduate Institute of Medical Education and Research, Chandigarh
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: INT/IEC/2016/937
Record Dates: First submitted 2017-04-06; First posted 2017-04-14 (Actual); Last update posted 2017-05-15 (Actual); Status verified 2017-04

CONDITIONS: Acid-Base Balance Disorder
MeSH Terms: interventions — Saline Solution; Plasmalyte A

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- normal saline (Experimental): Intravenous fluid used in these patients would be normal saline which would be given intravenously during intraoperative and postoperative period
  Interventions: Drug: intravenous fluid administration WITH NORMAL SALINE, PLASMALYTE A, OR RINGER LACTATE
- ringer lactate (Experimental): Intravenous fluid used in these patients would be ringer lactate which would be given intravenously during intraoperative and postoperative period
  Interventions: Drug: intravenous fluid administration WITH NORMAL SALINE, PLASMALYTE A, OR RINGER LACTATE
- plasmalyte A (Experimental): Intravenous fluid used in this arm in patients would be plasmalyte A which would be given intravenously during intraoperative and postoperative period
  Interventions: Drug: intravenous fluid administration WITH NORMAL SALINE, PLASMALYTE A, OR RINGER LACTATE

INTERVENTIONS:
Drug: intravenous fluid administration WITH NORMAL SALINE, PLASMALYTE A, OR RINGER LACTATE — intravenous fluid to be used for maintainance and replacement during renal transplant surgery will be normal saline, ringer lactate or plasmalyte A depending on the arm of intervention

SUMMARY:
Fluid management being an important component of surgery becomes more challenging for an anesthesiologist in case of renal transplant. Ischemia-reperfusion injury is an inevitable consequence of kidney transplantation, leading to metabolic acidosis .Normal saline (NS; 0.9% NaCl) is administered during kidney transplantation to avoid the risk of hyperkalemia associated with potassium-containing fluids. Plasmalyte is another fluid which can be used and probably will lead to better metabolic profile in these group of patients.The primary objective of this study will be to compare the effects of using normal saline (NS), Ringer lactate and Plasmalyte as intravenous fluids on acid-base balance and electrolytes during living donor kidney transplantation. Secondary outcomes assessed will be the effect on renal function.

ELIGIBILITY:
Inclusion Criteria:

* patients undergoing elective living donor renal transplant

Exclusion Criteria:

-

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 105 (Estimated)
Dates: Start 2015-04-01 (Actual); Primary Completion 2018-04 (Estimated); Study Completion 2018-04 (Estimated)

PRIMARY OUTCOMES:
acid base balance, 4 readings intraoperaively to be taken using arterial blood sample of the patient | during the surgery
  pH, pCO2, pO2, HCO3,Base deficit, Na, K are the values normally measured in acid base analysis

SECONDARY OUTCOMES:
serum creatinine on day 1, 2 and 7 of surgery | day 1, 2 and 7
  This is a function of kidney measure and will tell about the success of Renal Transplant
intraoperative hemodynamics in all patients | intraoperatively

CONTACTS AND LOCATIONS:
Locations (1):
- PGIMER, Chandigarh, India

IPD SHARING:
Plan to Share IPD: No